CLINICAL TRIAL: NCT03589040
Title: A Pharmacokinetic Evaluation of Etonogestrel Implant in HIV-infected Women on Darunavir Versus Ripilvirine-based Antiretroviral Therapy
Brief Title: Darunavir and Rilpivirine Interactions With Etonogestrel Contraceptive Implant
Acronym: DRIVE-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: University of Nebraska (Other); University of Pittsburgh (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Infectious Diseases Institute, Head of Department, Prevention Care and Treatment Infectious Diseases Institute, Makerere University College of Health Sciences, Makerere University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK21
Record Dates: First submitted 2018-05-28; First posted 2018-07-17 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: HIV; Contraception
MeSH Terms: interventions — etonogestrel; Drug Implants; Rilpivirine; Darunavir

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, open-label, parallel, two-group, sparse-sampling pharmacokinetic study to describe etonogestrel (ENG) pharmacokinetic parameters in two treatment groups (rilpivirine or darunavir- based antiretroviral therapy) in 60 HIV-1 infected women. The primary endpoint is the comparison of the mean ENG concentrations at month 6 between the rilpivirine or darunavir treatment groups versus historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ripivirine arm (Other): All subjects will be administered oral ripilvirine 25mg once daily together with the rest of their oral antiretroviral combination and an etonogestrel single-rod subdermal implant (68mg/rod). Study participants will have both interventions for a period of one year.
  Interventions: Drug: Etonogestrel 68Mg Implant; Drug: rilpivirine
- Darunavir arm (Other): All subjects will be administered oral DRV/r 600/100mg twice daily together with the rest of their oral antiretroviral combination and an etonogestrel single-rod subdermal implant (68mg/rod). Study participants will have both interventions for a period of one year.
  Interventions: Drug: Etonogestrel 68Mg Implant; Drug: darunavir

INTERVENTIONS:
Drug: Etonogestrel 68Mg Implant — Etonogestrel single-rod subdermal implant (68mg/rod) will be administered to all study participants
  Other Names: Implanon
Drug: rilpivirine — Oral rilpvirine 25mg
  Other Names: Edurant
  Arms: Ripivirine arm
Drug: darunavir — Oral darunavir+ritonavir 600/100mg
  Other Names: DRV
  Arms: Darunavir arm

SUMMARY:
This study will evaluate the pharmacokinetic properties of rilpivirine and darunavir when used in combination with etonogestrel

DETAILED DESCRIPTION:
Despite the benefits of hormonal contraceptives, significant drug-drug interactions (DDIs) with some antiretroviral therapies (ART) represent a barrier to effective family planning methods for HIV-infected women. It is therefore critical to generate data on the combined use of hormonal contraceptives and ART. This study is a prospective, non-randomized, open-label, parallel, two-group, sparse-sampling pharmacokinetic study to describe etonogestrel (ENG) pharmacokinetic (PK) parameters in two treatment groups (rilpivirine or darunavir- based ART) in 60 HIV-1 infected women. The primary endpoint is the comparison of the mean ENG concentrations at month 6 between the rilpivirine or darunavir treatment groups versus historical controls. This study will provide information on effective ART options for HIV positive women who opt for the contraceptive implant as a family planning method of choice.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Women age 18 years to 45 years
4. Diagnosed with HIV infection
5. Medically eligible for the ENG subdermal implant as a contraceptive method based on the WHO Medical Eligibility Criteria for Contraceptive Use
6. Receiving EFV- or LPV/r-based ART for a minimum of 1 year
7. If not abstinent, must agree to use an effective non-hormonal method of contraception for the duration of the study including male and female condoms or the copper-T intrauterine device.
8. Participants must have a negative urine pregnancy test at entry and report no unprotected sex since the last menstrual period or in the last two weeks.

   -

Exclusion Criteria:

1. HIV RNA greater than 50 copies/mL at the screening visit
2. CD4 count below 200 cells/mm3 at the screening visit
3. History of virologic failure on the current regimen (two consecutive viral load results equal to or greater than 400 copies/mL)
4. Serum hemoglobin less than 9.0 g/dl at screening
5. Elevations in serum levels of alanine transaminase (ALT) above 5 times the upper limit of normal
6. Elevations in serum creatinine above 2.5 times the upper limit of normal
7. Use of drugs known to be contraindicated with ENG, RPV (for women taking EFV-based ART), or DRV (for women taking LPV-based ART) within 30 days of study entry. Due to the dynamic nature of drug interactions related to antiretroviral therapy, the study team will review all concomitant medications at screening based on the US Department of Health and Human Services drug interaction table and the University of Liverpool HIV drug interaction tables (www.hiv-druginteractions.org)
8. Currently pregnant or postpartum <30 days at study entry.
9. Breastfeeding women within 6 months of delivery.
10. Patients with a history of hypersensitivity to ENG implant, undiagnosed vaginal bleeding, diagnosed or suspected sex hormone dependent neoplasia, benign or malignant liver tumor, or thromboembolic disease.
11. Presence of any active clinically significant disease or life-threatening disease that, in the investigator's opinion, would compromise the subject's safety or outcome of the study.

    -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of etonogestrel | Six months of combined use.
  Comparison of the mean etonogestrel concentrations at month 6 between rilpivirine and darunavir treatment groups versus historical controls.

SECONDARY OUTCOMES:
Concentration of rilpivirine and darunavir | 12 months
  Rilpivirine and darunavir mean concentration changes prior to implant placement and then over the duration of the study time period.
Number and severity of adverse events | 12 months
  Any signs and symptoms related to hormone exposure, including abnormal vaginal bleeding and local or systemic adverse events observed during the study period in both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Lamorde, PhD, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institue, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No